CLINICAL TRIAL: NCT02343445
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of P-1037 Solution for Inhalation in Patients With Cystic Fibrosis (CF)
Brief Title: Clearing Lungs With Epithelial Sodium Channel (ENaC) Inhibition in Cystic Fibrosis (CF)
Acronym: CLEAN-CF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS-G201
Record Dates: First submitted 2015-01-13; First posted 2015-01-22 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- P-1037 in Hypertonic Saline (HS) (Experimental): P-1037 Solution for Inhalation, 85 μg twice daily (BID) (28.3 μg/mL) in hypertonic saline (4.2% saline) BID
  Interventions: Drug: P-1037; Drug: Hypertonic Saline
- P-1037 in Saline (Experimental): P-1037 Solution for Inhalation, 85 μg BID (28.3 μg/mL) in 0.17% saline BID
  Interventions: Drug: P-1037; Drug: Saline
- Saline (Placebo Comparator): Placebo (0.17% saline) BID
  Interventions: Drug: Saline
- Hypertonic Saline (Sham Comparator): Hypertonic saline (4.2% saline) BID
  Interventions: Drug: Hypertonic Saline

INTERVENTIONS:
Drug: P-1037 — P-1037 is a novel ENaC inhibitor
  Arms: P-1037 in Hypertonic Saline (HS); P-1037 in Saline
Drug: Hypertonic Saline — 4.2% saline solution
  Arms: Hypertonic Saline; P-1037 in Hypertonic Saline (HS)
Drug: Saline — 0.17% saline solution
  Arms: P-1037 in Saline; Saline

SUMMARY:
The goal of the study is to evaluate the safety and tolerability of P-1037 and to determine whether the combination of P-1037 with hypertonic saline or P-1037 alone has a greater effect on lung function in patients with CF than placebo (0.17% saline).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 12 years of age or older.
* Diagnosis of cystic fibrosis as determined by the 1997 CF Consensus criteria (NIH Consensus Statement, 1997)
* Non-smoker
* FEV1 at Screening Visit 1 between 40% and 90%
* Stable regimen of CF medications and chest physiotherapy for the 28 days prior to Screening. Must be willing to discontinue use of hypertonic saline for the duration of the study.
* Clinically stable for at least 2 weeks
* All females of child-bearing potential must have a negative serum pregnancy test and if sexually active must agree to practice a highly effective form of contraception throughout the study and for 28 days after the last dose of study medication.

Exclusion Criteria:

* History of any organ transplantation or any significant disease or disorder
* Use of diuretics (including amiloride) or renin-angiotensin antihypertensive drugs or trimethoprim in the 28 days prior to Screening
* History of significant intolerance to inhaled hypertonic saline, as determined by the Investigator
* Known hypersensitivity to the study drug or amiloride
* Any clinically significant laboratory abnormalities at Screening Visit 1 as judged by the investigator, or any of the following:

  * Potassium ≥ 5 milliequivalent per Liter (mEq/L)
  * Abnormal renal function
  * Abnormal liver function, defined as ≥ 3 x upper limit of normal (ULN)
  * Hemoglobin level < 10.0 g/dL
* Female who is pregnant or lactating
* History of sputum or throat swab culture yielding Burkholderia species or Mycobacterium abscessus within 2 years of screening
* Has previously participated in an investigational trial involving administration of any investigational compound or use of an investigational device with 28 days prior to Screening
* Currently being treated with any ivacaftor containing regimen

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety (number of adverse events of P-1037 in treatment groups) | Day 15
  number of adverse events of P-1037 in treatment groups
Safety [change in forced expiratory volume in one second (FEV1) from predosing to 1 hour post dosing] | Day 1
  change in FEV1 from predosing to 1 hour post dosing with P-1037 in 4.2 % hypertonic saline and P-1037 in 0.17% saline

SECONDARY OUTCOMES:
Absolute change in FEV1 | Day 15
  change in FEV1, from baseline (immediately before first dose) to same time of day on Day 15
Effect of P-1037 on other forced vital capacity (FVC) measures (change in FVC from baseline (immediately before first dose) to same time of day on Day 15) | Day 15
  change in FVC from baseline (immediately before first dose) to same time of day on Day 15
Effect of P-1037 on Cystic Fibrosis Questionnaire - Revised (CFQ-R) | Day 15
  CFQ-R on Day 15
Determine whether co-administration of hypertonic saline (HS) enhances the effect of P-1037 on FEV1 (FEV1 on Day 15) | Day 15
  FEV1 on Day 15
Effect of P-1037 on (forced expiratory flow at 25%-75% of vital capacity (FEF25-75%) | Day 15
  FEF25-75% from baseline (immediately before first dose) to same time of day on Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Karl Donn, Study Chair — Parion Sciences
Locations (33):
- United States (33):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Univ of Florida Dept of Medicine, Gainesville, Florida
  - University of Miami Adult CF Center, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - New Lung Associates, Tampa, Florida
  - Chicago Cystic Fibrosis Institute, Glenview, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - UMass Memorial medical Center, Worcester, Massachusetts
  - Wayne State University/Harper University Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgets-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Pediatric Pulmonology/Cystic Fibrosis, Somerville, New Jersey
  - Albany Medical College, Albany, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Santiago Reyes, Oklahoma City, Oklahoma
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Anderson Pharmaceutical Research, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Children's Chest Associates, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - Univ of Texas Health Science Center, Tyler, Texas
  - University of Virginia Childrens, Charlottesville, Virginia
  - University of Wisconsin UW Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided